CLINICAL TRIAL: NCT02687282
Title: Ramathibodi Hospital, Mahidol University
Brief Title: Mallampati Score Before and After Cesarean Delivery
Acronym: MSBAC
Status: Completed | Type: Observational
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Lisa Sangkum, Principle investigator, Ramathibodi Hospital
Other Study IDs: Ramaanes2559
Record Dates: First submitted 2016-01-27; First posted 2016-02-22 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Alteration of Modified Mallampati Score
Keywords: Modified Mallampati score; Cesarean delivery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Evaluate upper airway changes — Evaluate upper airway changes at several point of time before and after cesarean delivery

SUMMARY:
Mallampati class change has not been well evaluated during the cesarean delivery. Various factors regarding to cesarean delivery might influence this changes. The aim of this study was to evaluate the Mallampati class before and after cesarean delivery and to identify predictive factors of the changes..

Study Type: Observational Cross-sectional study

DETAILED DESCRIPTION:
Mallampati class, thyromental distance, neck circumference, and upper lip bite test were evaluated at four time intervals : during pre-anesthetic visit (T0), 1-hour (T1), 6-hour (T2), and 24-hour after delivery (T3).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women scheduled for cesarean section, age ≥ 18 y at gestational age ≥ 37 weeks giving written informed consent.
* Initial Mallampati score ≤ III
* Normal clinical course

Exclusion Criteria:

* Patient who denied to participate the study
* Initial Mallampati score ≥ IV
* Age < 18 years old

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thai pregnant women scheduled for cesarean section, age ≥ 18 y at gestational age ≥ 37 weeks giving written informed consent.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluate Modified Mallampati score changes before and after cesarean delivery | up tp 2 days
  Modified Mallampati score (score 1-4;1= easy airway and 4 = difficult airway) before delivery, 2 and 6 hours after delivery, and post-operative day1 (the day of surgery and post-operative day 1)
Evaluate thyromental distance changes before and after cesarean delivery | up tp 2 days
  thyromental distance (centimeter) before delivery, 2 and 6 hours after delivery, and post-operative day1 (the day of surgery and post-operative day 1)
Evaluate upper lip bite score changes before and after cesarean delivery | up to 2 days
  Upper lip bite score (score 1-4; 1 = easy airway and 4 = difficult airway) before delivery, 2 and 6 hours after delivery, and post-operative day1 (the day of surgery and post-operative day 1)
Evaluate neck circumference changes before and after cesarean delivery | up to 2 days
  Neck circumference (centimeter) before delivery, 2 and 6 hours after delivery, and post-operative day1 (the day of surgery and post-operative day 1)

SECONDARY OUTCOMES:
Oxytocin dosage and Alteration of Modified mallampati score | up tp 2 days
  Evaluate the percentage of patients whose mallampati score increase from baseline between patient who recieved high dose oxytocin (≥ 0.6 U/minl) and low dose oxytocin ( <0.6 U/min )
Intraoperative intravenous fluid and Alteration of Modified mallampati score | up tp 2 days
  Evaluate the percentage of patients whose mallampati score increase from baseline between patient who recieved intravenous fluid ≥ 2000 ml and < 2000 ml
Estimate blood loss and Alteration of Modified mallampati score | up tp 2 days
  Evaluate the percentage of patients whose mallampati score increase from baseline between patient whose estimate blood loss≥ 1000 ml and < 1000 ml

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quinn AC, Milne D, Columb M, Gorton H, Knight M. Failed tracheal intubation in obstetric anaesthesia: 2 yr national case-control study in the UK. Br J Anaesth. 2013 Jan;110(1):74-80. doi: 10.1093/bja/aes320. Epub 2012 Sep 17. PMID 22986421
- [Background] Hawkins JL, Chang J, Palmer SK, Gibbs CP, Callaghan WM. Anesthesia-related maternal mortality in the United States: 1979-2002. Obstet Gynecol. 2011 Jan;117(1):69-74. doi: 10.1097/AOG.0b013e31820093a9. PMID 21173646
- [Background] Chang J, Streitman D. Physiologic adaptations to pregnancy. Neurol Clin. 2012 Aug;30(3):781-9. doi: 10.1016/j.ncl.2012.05.001. Epub 2012 Jun 30. PMID 22840789
- [Background] Kodali BS, Chandrasekhar S, Bulich LN, Topulos GP, Datta S. Airway changes during labor and delivery. Anesthesiology. 2008 Mar;108(3):357-62. doi: 10.1097/ALN.0b013e31816452d3. PMID 18292672
- [Background] Randell T. Prediction of difficult intubation. Acta Anaesthesiol Scand. 1996 Sep;40(8 Pt 2):1016-23. doi: 10.1111/j.1399-6576.1996.tb05620.x. PMID 8908216
- [Background] Rocke DA, Murray WB, Rout CC, Gouws E. Relative risk analysis of factors associated with difficult intubation in obstetric anesthesia. Anesthesiology. 1992 Jul;77(1):67-73. doi: 10.1097/00000542-199207000-00010. PMID 1610011
- [Background] Aydas AD, Basaranoglu G, Ozdemir H, Dooply SL, Muhammedoglu N, Kucuk S, Saidoglu L. Airway changes in pregnant women before and after delivery. Ir J Med Sci. 2015 Jun;184(2):431-3. doi: 10.1007/s11845-014-1138-8. Epub 2014 May 24. PMID 24859287
- [Background] Bhavani-Shankar K, Lynch EP, Datta S. Airway changes during Cesarean hysterectomy. Can J Anaesth. 2000 Apr;47(4):338-41. doi: 10.1007/BF03020949. PMID 10764179
- [Background] Boutonnet M, Faitot V, Katz A, Salomon L, Keita H. Mallampati class changes during pregnancy, labour, and after delivery: can these be predicted? Br J Anaesth. 2010 Jan;104(1):67-70. doi: 10.1093/bja/aep356. PMID 20007793
- [Background] Farcon EL, Kim MH, Marx GF. Changing Mallampati score during labour. Can J Anaesth. 1994 Jan;41(1):50-1. doi: 10.1007/BF03009661. PMID 8111943
- [Background] Guru R, Carere MD, Diwan S, Morau EL, Saunders J, Shorten GD. Effect of epidural analgesia on change in Mallampati class during labour. Anaesthesia. 2013 Jul;68(7):765-9. doi: 10.1111/anae.12288. Epub 2013 May 24. PMID 23710682
- [Background] Honarmand A, Safavi MR. Prediction of difficult laryngoscopy in obstetric patients scheduled for Caesarean delivery. Eur J Anaesthesiol. 2008 Sep;25(9):714-20. doi: 10.1017/S026502150800433X. Epub 2008 May 9. PMID 18471331
- [Background] Hu J, Huang S, Tian F, Sun S, Li N, Xie Y. A comparison of upper airway parameters in postpartum patients: vaginal delivery vs. caesarean section. Int J Clin Exp Med. 2014 Dec 15;7(12):5491-7. eCollection 2014. PMID 25664060
- [Background] Pilkington S, Carli F, Dakin MJ, Romney M, De Witt KA, Dore CJ, Cormack RS. Increase in Mallampati score during pregnancy. Br J Anaesth. 1995 Jun;74(6):638-42. doi: 10.1093/bja/74.6.638. PMID 7640115
- [Background] Ripolles Melchor J, Espinosa A, Martinez Hurtado E, Casans Frances R, Navarro Perez R, Abad Gurumeta A, Calvo Vecino JM. Colloids versus crystalloids in the prevention of hypotension induced by spinal anesthesia in elective cesarean section. A systematic review and meta-analysis. Minerva Anestesiol. 2015 Sep;81(9):1019-30. Epub 2014 Dec 11. PMID 25501602
- [Background] Idehen HO, Amadasun FE, Ekwere IT. Comparison of intravenous colloid and colloid-crystalloid combination in hypotension prophylaxis during spinal anesthesia for cesarean section. Niger J Clin Pract. 2014 May-Jun;17(3):309-13. doi: 10.4103/1119-3077.130231. PMID 24714008
- [Background] Baker P. Assessment before airway management. Anesthesiol Clin. 2015 Jun;33(2):257-78. doi: 10.1016/j.anclin.2015.02.001. PMID 25999001
- [Background] Hashim K, Thomas M. Sensitivity of palm print sign in prediction of difficult laryngoscopy in diabetes: A comparison with other airway indices. Indian J Anaesth. 2014 May;58(3):298-302. doi: 10.4103/0019-5049.135042. PMID 25024473